CLINICAL TRIAL: NCT05871294
Title: Cohort Study on Biomarkers and Clinical Treatment of Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhiwu Huang, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Zhiwu Huang, Ph.D., Professor, PHD, Director of the Hearing Center, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH9H-2022-T379-1
Record Dates: First submitted 2023-04-22; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Tinnitus, Subjective; Acoustic Stimulation; Transcranial Magnetic Stimulation, Repetitive; Magnetoencephalography
MeSH Terms: conditions — Tinnitus | interventions — Acoustic Stimulation; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acoustic stimulation therapy (Experimental): Patients in this group will receive acoustic stimulation therapy.
  Interventions: Device: Acoustic stimulation
- Repetitive transcranial magnetic stimulation therapy (Experimental): Patients in this group will receive repetitive transcranial magnetic stimulation therapy.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Acoustic stimulation — The sound used for treatment is selected based on the patient's tinnitus frequency and loudness. Patients receive 90 minutes of acoustic stimulation therapy every day (at least 5 days per week). The entire treatment period is 3 months.
  Arms: Acoustic stimulation therapy
Device: Repetitive transcranial magnetic stimulation — The course of repeated transcranial magnetic stimulation therapy is 4 weeks, with 5, 5, 4, and 3 treatments per week, each lasting 90 minutes (including rest time)
  Arms: Repetitive transcranial magnetic stimulation therapy

SUMMARY:
The goal of this clinical trial is to search for biomarkers in tinnitus patients in tinnitus patients and changes in biomarkers before and after treatment. The main questions it aims to answer are:

* What are the biomarkers of tinnitus patients？
* How do these biomarkers change during treatment and is there a good correlation with behavioral outcomes? Participants will be asked to complete audiological examination, tinnitus assessment, and magnetoencephalography examination, and they will receive sound therapy or repetitive transcranial magnetic stimulation therapy.

DETAILED DESCRIPTION:
This study aims to use magnetoencephalography (MEG) to collect the resting state responses before and after treatment in the control group, tinnitus patients in the acoustic stimulation treatment group, and rTMS treatment group. Firstly, compare the differences in power spectrum and brain functional connectivity indicators between tinnitus patients and normal control groups in different frequency bands, providing a theoretical basis for clinical diagnosis, precise positioning of tinnitus damaged areas, and understanding the pathogenesis of tinnitus; Secondly, compare the electrophysiological functional indicators of tinnitus patients before and after treatment to reveal whether the damaged brain network can gradually reshape after treatment, and whether network information can serve as potential biomarkers to indicate the degree of tinnitus recovery; Finally, compare the effectiveness differences between the two treatment methods, analyze their influencing factors, and provide guidance for frequency band precise intervention and rehabilitation of chronic tinnitus patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjective tinnitus lasting for more than 6 months, with a score of>36 of the Tinnitus Disability Inventory (THI)；
2. The otoscopy examination showed that the ear canal and eardrum were normal, and the tympanic impedance maps of both ears were Type A, indicating that language ability met the requirements of language testing

Exclusion Criteria:

1. Family or congenital deafness history, ototoxicity drug use history, otitis media patients, etc
2. Suffering from major physical diseases (sensory and motor disorders, neurological disorders, brain injuries, and other organic diseases) or mental disorders
3. The patient has aggressive behavior and an impulse to damage the device
4. Metal in the body (including orthodontics, dental implants), tattoos, and heart stent surgery
5. Having claustrophobia
6. Contraindications to magnetic resonance examination

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
THI | Baseline
  the scores of tinnitus handicap inventory（0-100）
THI | within 7 days of treatment completion
  the scores of tinnitus handicap inventory（0-100）
THI | follow-up for 1 month after treatment completion
  the scores of tinnitus handicap inventory（0-100）
VAS | Baseline
  Visual Analog Scale (VAS) is used to evaluate the loudness of tinnitus. The score range is 0-10
VAS | within 7 days of treatment completion
  Visual Analog Scale (VAS) is used to evaluate the loudness of tinnitus. The score range is 0-10
VAS | follow-up for 1 month after treatment completion
  Visual Analog Scale (VAS) is used to evaluate the loudness of tinnitus. The score range is 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwu Huang, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No